CLINICAL TRIAL: NCT04768062
Title: A Phase 3, Multi-center, Open-label Extension Study to Assess the Safety and Efficacy of Viltolarsen in Ambulant Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: Study to Assess the Safety and Efficacy of Viltolarsen in Ambulant Boys With DMD (RACER53-X)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS-065/NCNP-01-302
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — viltolarsen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Viltolarsen (Experimental): Patients amenable to exon 53 skipping will receive viltolarsen intravenous (IV) infusions, weekly, at 80 mg/kg for up to 96 weeks.
  Interventions: Drug: Viltolarsen

INTERVENTIONS:
Drug: Viltolarsen — Received during weekly intravenous infusions
  Other Names: NS-065/NCNP-01

SUMMARY:
This is a Phase 3, multi-center, open-label extension study in ambulant boys with DMD who have completed the 48-week treatment period of either viltolarsen or placebo in Study NS-065/NCNP-01-301.

DETAILED DESCRIPTION:
This Phase 3 study is a multi-center, open-label extension study in ambulant boys with DMD who have completed the 48-week treatment period of either viltolarsen or placebo in Study NS-065/NCNP-01-301. Patients will receive viltolarsen administered IV at weekly doses of 80 mg/kg.

Study NS-065/NCNP-01-302 will be comprised of a 96-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has completed the NS-065/NCNP-01-301 study;
2. Patient's parent(s) or legal guardian(s) has (have) provided written informed consent and Health Insurance Portability and Accountability Act authorization, where applicable, prior to any study-related procedures; patients will be asked to give written or verbal assent according to local requirements;
3. Patient and parent(s)/guardian(s) are willing and able to comply with scheduled visits, investigational product (IP) administration plan, and study procedures.

Exclusion Criteria:

1. Patient had an adverse event in Study NS-065/NCNP-01-301 that, in the opinion of the investigator and/or the sponsor, precludes safe use of viltolarsen for the patient in this study;
2. Patient had a treatment which was made for the purpose of dystrophin or dystrophin-related protein induction after completion of Study NS-065/NCNP-01-301;
3. Patient took any other investigational drug(s) during or after completion of Study NS-065/NCNP-01-301;
4. Patient is judged by the investigator and/or the sponsor not to be appropriate to participate in the extension study for any reason.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related Adverse Events as assessed by CTCAE v4.03 | baseline to up to 96 weeks of treatment

SECONDARY OUTCOMES:
Time to Stand Test (TTSTAND) | baseline to 96 weeks of treatment
  Change in Time to Stand
Time to Run/Walk 10 Meters Test (TTRW) | baseline to 96 weeks of treatment
  Change in Time to Run/Walk 10 meters
Six-minute Walk Test (6MWT) | baseline to 96 weeks of treatment
  Change in Six-minute Walk
North Star Ambulatory Assessment (NSAA) | baseline to 96 weeks of treatment
  Change in North Star Ambulatory Assessment
Time to Climb 4 Stairs Test (TTCLIMB) | baseline to 96 weeks of treatment
  Change in Time to Climb 4 Stairs
Muscle Strength Measured by Hand-Held Dynamometer | baseline to 96 weeks of treatment
  Change in Muscle Strength Measured by Hand-Held Dynamometer

CONTACTS AND LOCATIONS:
Locations (31):
- Australia (2):
  - Queensland Children's Hospital, Brisbane
  - The Childrens Hospital at Westmead, Westmead
- CHU de Quebec Research Centre, Québec, Canada
- Chile (2):
  - Hospital de Niños Roberto del Rio, Santiago
  - Pontificia Universidad Católica de Chile, Santiago
- China (4):
  - Chinese PLA General Hospital, Beijing
  - Hunan Children's Hospital, Changsha
  - Children's Hospital of Fudan University, Shanghai
  - Shenzhen Children's Hospital, Shenzhen
- Fakultni nemocnice Hradec Kralove, Nový Hradec Králové, Czechia
- Greece (2):
  - Agia Sofia Children's Hospital, Athens
  - Hippokration General Hospital of Thessaloniki, Thessaloniki
- Fondazione Policlinico Universitario A. Gemelli - Universita Cattolica del Sacro Cuore, Rome, Italy
- National Center of Neurology and Psychiatry, Tokyo, Japan
- Instituto Nacional de Pediatría, Mexico City, Mexico
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen
- New Zealand Clinical Research Ltd., Auckland, New Zealand
- Rikshospitalet, Oslo, Norway
- Russia (3):
  - Russian National Research Medical University, Moscow
  - "Saint Petersburg State Paediatric Medical University" based at Consultative and Diagnostic Centre, Saint Petersburg
  - Tomsk National Research Medical Center of Russian Academy of Sciences, Tomsk
- South Korea (2):
  - Pusan National University Yangsan Hospital, Pusan
  - Seoul National University Hospital, Seoul
- Spain (2):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario La Paz, Madrid
- Yeditepe University Kosuyolu Hospital, Istanbul, Turkey (Türkiye)
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Hospital for Children, Glasgow
  - Royal Manchester Children's Hospital, Glasgow
  - University College London Institute of Child Health, London

REFERENCES:
- See also: Study to Assess the Efficacy and Safety of Viltolarsen in Ambulant Boys With DMD (RACER53) — https://clinicaltrials.gov/ct2/show/NCT04060199